CLINICAL TRIAL: NCT01570946
Title: A Pragmatic and Scalable Strategy Using Mobile Technology to Promote Sustained Lifestyle Changes to Prevent Type 2 Diabetes in India and the UK
Brief Title: Use of Mobile Technology to Promote Sustained Lifestyle Changes to Prevent Type 2 Diabetes in India and the UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Collaborators: Indian Council of Medical Research (Other Government); Medical Research Council (Other Government); Imperial College London (Other)
Responsible Party: Principal Investigator, Dr.A.Ramachandran, President, India Diabetes Research Foundation, India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 58/1/MRC-ICMR/09/NCD-II_018
Record Dates: First submitted 2012-03-03; First posted 2012-04-04 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Prediabetic State
Keywords: Lifestyle changes to prevent type 2 diabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle modification (Experimental): The mobile phone based intervention will use short messaging service (SMS or text messaging) to deliver education, treatment targets, advice, support and motivation.
  Interventions: Behavioral: Lifestyle Modification
- Standard Care (No Intervention): Baseline 30-minute interview delivering personalised diet and exercise advice supplemented with educational material on diabetes.

INTERVENTIONS:
Behavioral: Lifestyle Modification — The mobile phone based intervention will use short messaging service (SMS or text messaging) to deliver education, treatment targets, advice, support and motivation.
  Arms: Lifestyle modification

SUMMARY:
Primary prevention of diabetes is of paramount importance in both developed and in developing countries. Several studies including the Indian Diabetes Prevention Programmes have shown that Lifestyle modification in people with prediabetes can reduce the progression to diabetes by 58%. However, there are two main problems in applying diabetes prevention strategies to the population as a whole. (1) Trial based interventions are unrealistic on a population level in any country. (2) The oral glucose tolerance test applied so far to identify those at high risk is a poorly reproducible and time consuming test both for the participant and for health care workers. Hence more practical means of defining individuals who would benefit from lifestyle intervention are required.

The current study proposes a prevention strategy that will employ a lifestyle modification programme delivered by text messaging in both India and the UK.Subjects will be identified based on the HbA1c measurement instead of the oral glucose tolerance test. The study will also assess the efficacy, acceptability and cost effectiveness of mobile phone based intervention both in India and the UK.

Messages will be based to deliver education, treatment targets, advice, support and motivation. Subjects will be invited to participate and, once recruited, will be randomised to usual care or the SMS intervention group.

Usual care will consist of a one-to-one 30 minute interview, conducted by the research team, delivering personalised diet and exercise advice.

The intervention group will undergo the same initial interview and, in addition, will receive 3 times weekly text messaging with education, advice, support and motivation. These messages will be personalised to individual targets set at the initial interview.

Primary Outcome:Progression to Diabetes Secondary Outcomes will be based on Physical activity / Cardiovascular risk factors/and quality of life.

The study programme is compatible with major initiatives in both the UK and India for the prevention of diabetes and cardiovascular disease (CVD).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with no history of diabetes
* Persons with 2 or more risk factors including

  1. Age 35-55 years
  2. Positive family history of diabetes
  3. Body mass index ≥23kg/m2
  4. Waist circumference >90cm for men and >80cm for women
  5. Hypertension
  6. Sedentary habits
* HbA1c 6.0% - <6.5%

Exclusion Criteria:

* Known diabetes
* Any other illness
* Unwilling to participate

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1171 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Progression to diabetes | Participants will be assessed at 12-month, 24-month intervals from the time of randomisation for 2 years.
  The primary outcome is progression to diabetes assessed by HbA1c ≥6.5%.

SECONDARY OUTCOMES:
Improvements in physical activity | Participants will be assessed at 6 month intervals for 2 years.
  Improvement in physical activity defined as minutes per day of moderate-to-vigorous physical activity (MVPA) measured by Actigraph, total and domain-specific physical activity measured by Recent Physical Activity Questionnaire (RPAQ).
Improvements in cardiovascular risk factors | Participants will be assessed at 6-month, 12-month and 24-month intervals for 2 years.
  Measurement of insulin and lipid levels
Improvements in Quality of Life | Participants will be assessed at 12-month and 24-month intervals for 2 years.
  Quality of life measured by EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Ramachandran Ambady, MD., Ph.D., D.Sc., FRCP, Principal Investigator — President; Desmond G Johnston, MB ChB.,PhD.,FRCP.,FRCPath, Principal Investigator — Campus Dean, Imperial College London,Director, UK Diabetes Research Network; Nicholas J Wareham, MBBS.,M.Sc.Ph.D, Principal Investigator — Director, MRC Epidemiology Unit and co-Director Institute of Metabolic Science, University of Cambridge
Locations (2):
- India Diabetes Research Foundation, Chennai, Tamil Nadu, India
- Imperial College, London, United Kingdom

REFERENCES:
- [Background] Ramachandran A, Snehalatha C, Samith Shetty A, Nanditha A. Predictive value of HbA1c for incident diabetes among subjects with impaired glucose tolerance--analysis of the Indian Diabetes Prevention Programmes. Diabet Med. 2012 Jan;29(1):94-8. doi: 10.1111/j.1464-5491.2011.03392.x. PMID 21790773
- [Background] Shetty AS, Chamukuttan S, Nanditha A, Raj RK, Ramachandran A. Reinforcement of adherence to prescription recommendations in Asian Indian diabetes patients using short message service (SMS)--a pilot study. J Assoc Physicians India. 2011 Nov;59:711-4. PMID 22616337
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Background] Ramachandran A, Snehalatha C, Mary S, Selvam S, Kumar CK, Seeli AC, Shetty AS. Pioglitazone does not enhance the effectiveness of lifestyle modification in preventing conversion of impaired glucose tolerance to diabetes in Asian Indians: results of the Indian Diabetes Prevention Programme-2 (IDPP-2). Diabetologia. 2009 Jun;52(6):1019-26. doi: 10.1007/s00125-009-1315-x. Epub 2009 Mar 10. PMID 19277602
- [Background] Ramachandran A, Snehalatha C, Yamuna A, Mary S, Ping Z. Cost-effectiveness of the interventions in the primary prevention of diabetes among Asian Indians: within-trial results of the Indian Diabetes Prevention Programme (IDPP). Diabetes Care. 2007 Oct;30(10):2548-52. doi: 10.2337/dc07-0150. Epub 2007 Aug 1. PMID 17670917
- [Background] Ramachandran A, Riddle MC, Kabali C, Gerstein HC; ORIGIN Investigators. Relationship between A1C and fasting plasma glucose in dysglycemia or type 2 diabetes: an analysis of baseline data from the ORIGIN trial. Diabetes Care. 2012 Apr;35(4):749-53. doi: 10.2337/dc11-1918. Epub 2012 Feb 8. PMID 22323416
- [Derived] Nanditha A, Thomson H, Susairaj P, Srivanichakorn W, Oliver N, Godsland IF, Majeed A, Darzi A, Satheesh K, Simon M, Raghavan A, Vinitha R, Snehalatha C, Westgate K, Brage S, Sharp SJ, Wareham NJ, Johnston DG, Ramachandran A. A pragmatic and scalable strategy using mobile technology to promote sustained lifestyle changes to prevent type 2 diabetes in India and the UK: a randomised controlled trial. Diabetologia. 2020 Mar;63(3):486-496. doi: 10.1007/s00125-019-05061-y. Epub 2020 Jan 9. PMID 31919539
- [Derived] Thomson H, Oliver N, Godsland IF, Darzi A, Srivanichakorn W, Majeed A, Johnston DG, Nanditha A, Snehalatha C, Raghavan A, Susairaj P, Simon M, Satheesh K, Ramachandran A, Sharp S, Westgate K, Brage S, Wareham N. Protocol for a clinical trial of text messaging in addition to standard care versus standard care alone in prevention of type 2 diabetes through lifestyle modification in India and the UK. BMC Endocr Disord. 2018 Sep 10;18(1):63. doi: 10.1186/s12902-018-0293-8. PMID 30200935